CLINICAL TRIAL: NCT00944684
Title: Prospective, Open-label, Randomised Controlled Trial on Efficacy and Tolerability of PegIFN-alpha 2a + Serum Level-adapted RBV vs. PegIFN-alpha 2a + Weight-based RBV in Treatment-naive Patients With Chronic Hepatitis C Genotype 1
Brief Title: High Dose Ribavirin in the Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Roche Pharma AG (Industry); University of Lausanne (Other); Cantonal Hospital of St. Gallen (Other); Waid City Hospital, Zurich (Other); University of Basel (Other)
Responsible Party: Felix Stickel, University of Bern, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091/07; ML21071; SASL-24
Record Dates: First submitted 2009-07-17; First posted 2009-07-23 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Antiviral treatment; Ribavirin; Sustained virological response; Hemolytic anemia; Erythropoetin
MeSH Terms: conditions — Hepatitis C, Chronic; Anemia, Hemolytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): PegIFN-alpha 2a + RBV (commenced according to kidney function) adjusted to plasma levels. Treatment with erythropoetin 3x3,000IU/week up to 3x10,000IU/week in case of hemolytic anemia
  Interventions: Drug: High ribavirin dose
- B (Active Comparator): PegIFN-alpha 2a + RBV (weight based; 1,000 or 1,200 mg/day)
  Interventions: Drug: Standard ribavirin dose

INTERVENTIONS:
Drug: High ribavirin dose — Ribavirin dose started according to kidney function (usually 1,800mg) and adapted according to plasma level during follow-up
  Arms: A
Drug: Standard ribavirin dose — Ribavirin dose started at 1,000mg (body weight <65kg) or 1,200mg (body weight equal or >65kg)
  Arms: B

SUMMARY:
Treatment of patients with chronic hepatitis C infected with genotype 1 hepatitis C virus (HCV) consists of combined peginterferon/ribavirin for 48 weeks. Approximately 50% of patients experience sustained virological response which equals cure. All other patients either do not respond or experience recurrence of HCV virus and chronic hepatitis. Important predictors of successful treatment are sustained dosing of both peginterferon and ribavirin. With regard to the latter, clinical evidence indicates that higher ribavirin doses may in fact even improve treatment outcome. However, high ribavirin doses cause hemolytic anemia which require dose reductions. Recent clinical experience show that erythropoetic growth factors, including erythropoetin, can counteract hemolytic anemia caused by antiviral treatment in chronic hepatitis C patients. Therefore, the current trial aims to test whether higher ribavirin doses adapted to a target plasma concentrations instead of a weight-based dosing result in better healing rates, and whether ribavirin-associated hemolytic anemia can be compensated by concommitant erythropoetin treatment.

Using a randomized, controlled, open-label design, the investigators hypothesize that patients with high ribavirin doses adapted to plasma levels experience better viral clearance than patients treated with standard weight-based ribavirin doses. In addition, the investigators hypothesize that erythropoetin treatment will counteract hemolytic anemia induced by ribavirin thereby allowing maintenance of target plasma concentrations without ribavirin dose reductions.

DETAILED DESCRIPTION:
Background

Prevalence and incidence of chronic hepatitis C (CHC) are rising worldwide. Complications include chronic liver failure and hepatocellular carcinoma, and chronic hepatitis C is a major indication for liver transplantation. Effective treatment is required to prevent these outcomes.

Current treatment consists of a combination of peginterferon (PegIFN) and ribavirin (RBV) given for 24 or 48 weeks depending on the viral genotype. While genotypes 2 and 3 respond well to 24 weeks of PegIFN/RBV with approximately 80% viral clearance, genotype 1 infected patients only achieve about 40-50% sustained viral response (SVR) with 48 weeks of combination therapy.

RBV is a nucleoside analog with structural similarities to guanosine, which modulates RNA and DNA synthesis. RBV reveals antiviral activity against respiratory syncytial (RS)-virus, influenza virus, Lassa virus uand others. The exact mode of antiviral activity is yet unknown but believed to relate to reducing survival of HCV-infected hepatocytes thereby allowing for elimination of infected cells by interferon-stimulated immune mechanisms.

Generally, RBV is well tolerated. With standard daily doses between 1.000 and 1.200mg, irritability, sleeping abnormalities, cough and pruritus. The most prevalent and typical side effect of RBV is a dose-dependent hemolytical anemia which responds well to dose reduction or interruption of RBV therapy. RBV-associated anemia impairs quality of life and, overall, 25-36% of patients require dose reductions and/or RBV cessation. However, reduction/cessation of RBV is associated with a significant drop of SVR and measures to maintain RBV doses are clearly warranted. Several recent studies have shown that erythropoetin can counteract RBV-induced hemolytic anemia, and improve quality of life.

The relevance of RBV dose with regard to therapeutic response to combination therapy is well-established and currently, RBV is dosed according to weight: patients with CHC genotype 1 are treated with 1.000mg if body weight is <65kg, and receive 1.200mg if >65kg.

Retrospective studies have shown that relapsers and non-responders to antiviral treatment with RBV had lower RBV levels than those who had a SVR. In a retrospective analysis of 4 studies investigating a total of 1105 patients treated with RBV, RBV plasma concentrations measured at 4 weeks of treatment correlated with viral clearance: SVR was 31.8% in those with RBV levels <1,000ng/ml, and increased to 62.5% with RBV concentrations at >4,000ng/ml.

A pilot trial from Sweden investigated whether dosing RBV according to a plasma level of 15mcmol/l (3.7mcg/ml) in 10 patients. Median RBV dose was 2.540mg/day and all patients received erythropoetin.SVR was achieved in 9 of 10 patients.

So far, a randomized, controlled trial comparing weight-based RBV (standard) vs. RBV dosed according to kidney function and plasma levels.

Objective

Comparison of efficacy and tolerability of treatment with PegIFN-alpha 2a + RBV dosed according plasma concentrations vs PegIFN-alpha 2a + weight-based RBV in patients with chronic hepatitis C genotype 1

Methods

Prospective, controlled, open label randomized human trial

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years
* Elevated liver enzymes levels
* Compensated liver disease
* Available liver histology confirming METAVIR F2 fibrosis
* Written consent to participation

Exclusion Criteria

* Age <18, >65
* Prior ribavirin treatment
* Intolerance towards ribavirin, PegIFN or erythropoetin
* Pregnancy or breast feeding
* Relevant cardiovascular or pulmonary disease
* Kidney insufficiency (creatinine clearance <50ml/min)
* Coinfection with HIV or hepatitis B virus
* Hepatic comorbidities (hemochromatosis, Wilson's disease, autoimmune disorders)
* Alcohol consumption > 40g/day
* Psychiatric disorders
* Malignancy (except for basalioma)
* Active consumption of illicit drugs
* Participation in another trial shorter than 3 months prior to inclusion
* Lack of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 1 Day

SECONDARY OUTCOMES:
Adverse Events | day 1 until 24 weeks after end or treatment
Rapid virological response at 4 weeks of treatment | 4 weeks
Early virological response at 12 weeks of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Felix Stickel, MD, Principal Investigator — Institute for Clinical Pharmacology and Visceral Research, University of Bern
Locations (5):
- Switzerland (5):
  - Dept of Gastroenterology, University of Basel, Basel
  - Institute of Clinical Pharmacology and Visceral Research, University of Bern, Bern
  - Division of Gastroenterology, University of Lausanne, Lausanne
  - Kantonsspital St.Gallen, Sankt Gallen
  - Stadtspital Waid, Zürich, Zurich

REFERENCES:
- [Derived] Pfaundler N, Kessebohm K, Blum R, Stieger M, Stickel F. Adding pancreatic panniculitis to the panel of skin lesions associated with triple therapy of chronic hepatitis C. Liver Int. 2013 Apr;33(4):648-9. doi: 10.1111/liv.12119. Epub 2013 Feb 15. No abstract available. PMID 23410147